CLINICAL TRIAL: NCT04948112
Title: Effectiveness of Real-time Continuous Glucose Monitoring (CGMS) to Improve Glycemic Control in Patients with Early Gestational Diabetes Mellitus: a Randomized Controlled Trial Using CGMS Vs. Self-monitoring Blood Glucose (SMBG)
Brief Title: Effectiveness of CGMS Vs. Self-monitoring Blood Glucose (SMBG) in Woman with Gestational Diabetes
Acronym: STEADYSUGAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woman's (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RP-21-012
Record Dates: First submitted 2021-06-22; First posted 2021-07-01 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: continuous glucose monitoring

STUDY DESIGN:
Intervention Model Description: Randomized control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Real-time (rt) CGMS with SMBG (Experimental): Real time continuous glucose monitoring plus self-monitored blood glucose
  Interventions: Device: real time continuous glucose monitor
- SMBG with blinded CGM (Active Comparator): Self monitored blood glucose with blinded continuous glucose monitoring
  Interventions: Device: blinded continuous glucose monitor

INTERVENTIONS:
Device: real time continuous glucose monitor — CGM sensor will read blood glucose every 10 minutes
  Other Names: Dexcom G6
  Arms: Real-time (rt) CGMS with SMBG
Device: blinded continuous glucose monitor — CGM that records blood glucose but not visible to patient
  Other Names: blinded Dexcom
  Arms: SMBG with blinded CGM

SUMMARY:
The detection of and control of gestational diabetes carries benefits for both mother and baby related to immediate pregnancy outcomes. The glycemic disorders in diabetes are not solely limited to fasting and postprandial hyperglycemia, but can be extended to the glycemic variability that includes both upward (postprandial glucose increments) and downward (interprandial glucose decrements) changes. Glycemic variability, as a component of the glycemic disorders, has more deleterious effects than sustained chronic hyperglycemia in the development of diabetic complications. Glycemic variability is associated with increased risks of adverse pregnancy outcomes in GDM. Hyperglycemic excursion has been shown to be the strongest predictor of macrosomia, the most common complication of pregnancy with diabetes. When compared with routine standard antenatal care, continuous glucose monitoring system (CGMS) guided treatments should signiﬁcantly improve glycemic control, lower infant birth weight, and reduce risk of macrosomia in gestational women with diabetes. We will investigate the following questions (1) Whether CGMS can detect greater glycemic variability in women with an early GDM diagnosis; (2) Whether CGMS can subsequently moderate treatment strategies of GDM especially patient behavior and glucose levels; (3) Whether CGMS can eventually improve maternal (i.e., reduce gestational weight gain and lower glycemic levels during pregnancy) and fetal outcomes (reduce LGA babies and C-section rate) compared with traditional self-monitored blood glucose (SMBG) use.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is defined as any degree of glucose intolerance with onset during pregnancy. It is associated with increased feto-maternal morbidity as well as with long-term complications in the mother and offspring . GDM is associated with significant complications during pregnancy, including an increased need for Cesarean sections; higher risks of ketonemia, preeclampsia, and urinary tract infection in both mothers and infants; increased perinatal morbidity (e.g., macrosomia, neonatal hypoglycemia, and neonatal jaundice); and possibly mortality. The risk of complications in women with GDM increases proportionally with the worsening of glycemic tolerance. Comprehensive glucose monitoring and therapy are indispensable to prevent these complications because even small increases in maternal glucose are related to poorer clinical outcomes. Treatment of GDM during pregnancy, centers on dietary modulation, promotion of healthy physical activity and pharmacologic management, primarily with insulin as well as oral hypoglycemic agents (OHA), if glycemic control cannot be achieved with lifestyle measures alone. The details of the therapeutic approach, in particular regarding various dietary approaches and the potential use of OHAs such as metformin and glyburide (glibenclamide) differ widely between and within countries. Two landmark prospective randomized controlled trials have confirmed that detection of and control of GDM carries benefits for both mother and baby in terms of immediate pregnancy outcomes. Women in the intervention arm of the Australian (Crowther) study showed lower rates of fetal macrosomia, reduced frequency of large-for-gestational age (LGA) babies and reduced preeclampsia. In the US (Landon) study, women who received treatment for GDM demonstrated lower gestational weight gain (GWG) and lower rates of pre-eclampsia. Reduced frequency of LGA and macrosomia were noted in infants of treated mothers.

Glucose monitoring targets in pregnancy need to be tight, with low thresholds for commencing pharmacotherapy or increasing the insulin dosage. The Hyperglycemia and Adverse Pregnancy Outcomes (HAPO) study showed that a fasting glucose of 5.1 mmol/L in the oral glucose tolerance test at 24-28 weeks of gestation was already associated with a 75% increased risk of adverse outcomes . Self monitoring of blood glucose (SMBG) is a frequently used method to monitor blood glucose during pregnancy. However, this method is not sufficient to detect all glycemic fluctuations. Since the initiation of insulin/metformin/glyburide therapy and the related dosage adjustments depend solely on the SMBG results, inaccurate results may lead to a greater chance of hypo- or hyperglycemia and may even fail to detect hypoglycemic episodes. Therefore, accurate SMBG results are crucial for management of hyperglycemia during pregnancy. The capabilities of continuous glucose monitoring systems (CGMS) during pregnancy have advanced with the technical aspects of glucose meters, and therefore considering these aspects is important during pregnancy. Continuous glucose monitoring (CGM) provides unique insights into daily glycemic control and permits a better understanding of how glucose variability may influence acute and long-term complications of diabetes. Real-time CGM by providing glucose measurements as often as every 5 minutes, low and high glucose alerts, and glucose trend information, has the potential to better inform diabetes management decisions compared with episodic self-monitoring with a SMBG. CGM offers a potential source of data required to improve the detection and management of glucose levels in diabetic pregnancy. CGM provides far more frequent glucose measurements than SMBG and far more information on short-to-medium-term trends in glucose levels than either SMBG or even HbA1c. The slow kinetics of glycosylated hemoglobin accumulation and physiological changes in erythrocyte formation during pregnancy mean that A1C is only a limited predictor of acute blood glucose changes providing an explanation for the poor pregnancy outcomes, even in women with apparently "good" glycemic control . Recent attention has therefore focused on evaluating the role of CGMS in pregnancy with studies providing normative data in diabetic and nondiabetic pregnancies. CGMS is also capable of recording glucose levels throughout both day and night without disrupting the normal activities of daily living (particularly periods of activity, rest, and sleep). A real time-CGMS provides the patient with continuous information about the alterations in the blood glucose levels throughout the day, which is immediately revealed to the patient, and helps the patient to understand how food, exercise, and insulin affect blood glucose. This visibility may empower the patient to modify his/her lifestyle and engage in therapeutic management. CGMS data allows us to better understand where, when, and how we might better invest our efforts to optimize glucose control in diabetic pregnancy to reduce LGA and improve pregnancy outcomes.

CGMS use has been successful, safe, and accurate in detecting glucose levels in pregnancies with diabetes. RT-CGMS studies in non-pregnant type 1 and type 2 diabetes patients reported its efficacy in improving glycemic control. The effectiveness of CGMS in improving pregnancy outcomes complicated by GDM is still understudied. In a study by Wei and colleagues, a total of 106 women with GDM in gestational weeks 24-28 were randomly allocated to the antenatal care plus CGMS group or the self-monitoring blood glucose (SMBG) group. The CGMS group was subdivided into early and late subgroups. There were no significant differences in prenatal or obstetric outcomes, e.g., caesarean delivery rate, Apgar score at 5 min, macrosomia or neonatal hypoglycemia, between the CGMS and SMBG groups. The CGMS group had lower glycated hemoglobin (HbA1C) levels than the SMBG group; however, the difference was not statistically significant. The proportion of GDM women with excessive gestational weight gain was lower in the CGMS group than in the SMBG group (33.3% vs. 56.4%, P = 0.039), and women who initiated CGMS earlier gained less weight (P = 0.017). The mode of blood glucose monitoring (adjusted OR 2.40; 95% CI 1.030-5.588; P = 0.042) and pre-pregnancy BMI (adjusted OR 0.578; 95% CI 0.419-0.798; P = 0.001) were independent factors for weight gain. The investigators concluded that early CGMS for GDM mothers reduced gestational weight gain. Voormolen et al. randomized 109 women with GDM to CGMS vs. standard treatment (SMBG 4-8 times daily and HbA1c levels every 4 weeks). Compared with SMBG users, CGMS users had a significantly lower incidence of pre-eclampsia [Relative Risk (RR) 0.3; 95%Cl: 0.12-0.8]. In another study, Yu et al. recruited 340 women with GDM and assigned 190 to routine care (SMBG 7 times daily) and the other 150 to 72 h CGMS. Compared with SMBG, CGMS users tended to have lower incidence of pre-eclampsia [5out of 150 (3.3%) vs. 19 out of 190 (10%), P = 0.019], primary cesarean section [51 out of 150 (34.0%) vs. 88 out of 190 (46.3%), P =0.028], and premature delivery [7 out of 150 (4.7%) vs. 22 out of 190 (11.6%), P = 0.024]. In addition, intermittent use of retrospective CGM in pregnant women with pre-gestational diabetes or GDM was associated with improvement in blood glucose and pregnancy outcomes.

This is a randomized controlled trial (RCT) which will assess CGMS vs. SMBG by allowing all participants to use both methods but the SMBG group will be blinded to CGMS. A total of 121 women with gestational diabetes mellitus (GDM) diagnosed in gestational weeks 8-25 (6+0 to 25+6weeks) (by 8 weeks we can detect heartbeat and consider it a viable pregnancy) will be recruited. We will investigate the following questions (1) Whether CGMS can detect greater glycemic variability in women with an early GDM diagnosis; (2) Whether CGMS can subsequently moderate treatment strategies of GDM especially patient behavior and glucose levels; (3) Whether CGMS can eventually improve maternal (i.e., reduce gestational weight gain and lower glycemic levels during pregnancy) and fetal outcomes (reduce LGA babies and C-section rate) compared with traditional SMBG use.

ELIGIBILITY:
Inclusion Criteria:

* • 8-26 weeks gestation

  * singleton pregnancy,
  * a positive oral glucose tolerance test
  * written informed consent.

Exclusion Criteria:

* • prior diagnosis of diabetes mellitus,

  * presence of infection,
  * Presence of significant systemic disease or other severe metabolic, endocrine, medical co-morbidities
  * history of bariatric surgery or other surgeries that induce malabsorption
  * long-term use (>2 weeks) of systemic steroids prior to enrolment
  * multiple pregnancy
  * patients already using glucose lowering medications (metformin or insulin) before study entry
  * fetal growth restriction due to placental dysfunction at study entry
  * History of major depressive or other severe psychiatric disorders or inpatient psychiatric treatment up to 1year before enrolment
  * Inability or refusal to comply with protocol
  * Currently participating or having participated in an experimental study in previous three months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — must be pregnant
Enrollment: 128 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Average percent time in glucose range | up to 32 weeks
  average time in hours and minutes spent in target glucose range

SECONDARY OUTCOMES:
time spent in hyperglycemia (time above range) | up to 32 weeks
  average time in hours and minutes spent with elevated blood glucose
time spent in hypoglycemia (time below range) | up to 32 weeks
  average time in hours and minutes spent with low blood glucose
percent weight gain during pregnancy | through study completion, an average of 38 weeks
  change in bodyweight during pregnancy
HbA1c | through study completion, an average of 38 weeks
  change (lowering or increasing) HbA1C
Large-for -gestational age newborns | at time of delivery
  the proportion of LGA newborns (birth weight >90th percentile)
Neonatal hypoglycemia | at time of delivery
  blood glucose level below 2.2 mmol/L (40 mg/dL)

OTHER OUTCOMES:
CGM-satisfaction (CGM SAT) survey | immediately after delivery
  survey of how satisfied the subject is with their CGM (real time CGM only)
Perceived benefit questionnaire (GMS) | immediately after delivery
  participants satisfaction with and therapeutic impact of the glucose monitoring systems

CONTACTS AND LOCATIONS:
Overall Officials: Karen Elkind-Hirsch, PhD, Principal Investigator — Woman's Hospital, Louisiana
Locations (1):
- Karen Elkind-Hirsch, Baton Rouge, Louisiana, United States